CLINICAL TRIAL: NCT03632330
Title: SEDATION OF ADULT PATIENTS UNDERGOING GASTROINTESTINAL ENDOSCOPY: A NETWORK META-ANALYSIS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C0801043
Record Dates: First submitted 2018-07-30; First posted 2018-08-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2019-07

CONDITIONS: Gastrointestinal Endoscopy; Sedation; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Propofol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (4):
- Dexmedetomidine: Dexmedetomidine group
  Interventions: Drug: Dexmedetomidine
- Midazolam: Midazolam group
  Interventions: Drug: Midazolam
- propofol: propofol group
  Interventions: Drug: Propofol
- Midazolam/Propofol: Midazolam and Propofol group
  Interventions: Drug: Midazolam/Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine group
  Other Names: The group includes patients treated with Dexmedetomidine
  Groups: Dexmedetomidine
Drug: Midazolam — Midazolam group
  Other Names: The group includes patients treated with Midazolam
  Groups: Midazolam
Drug: Propofol — Propofol group
  Other Names: The group includes patients treated with Propofol
  Groups: propofol
Drug: Midazolam/Propofol — Midazolam/Propofol group
  Other Names: The group includes patients treated with Midazolam and propofol
  Groups: Midazolam/Propofol

SUMMARY:
The objective of this study is to compare the efficacy and safety of dexmedetomidine with other sedatives in sedation during endoscopy by analyzing the most recently published interventional trials and observational studies.

DETAILED DESCRIPTION:
A variety of sedatives are available in procedural sedation and the efficacy & safety have been compared in several trials for procedural sedation. However, none of clinical trial has enough number of patients to clarify the conclusive differences among sedatives. Thus, pooling all available studies together systematically by network meta-analysis for GI endoscopic procedure may provide a better understanding of efficacy and safety of sedatives. Therefore we would like to conduct a network meta-analysis to analyze the outcomes of GI endoscopy by using the most recently-published interventional trials.

ELIGIBILITY:
* Inclusion criteria We will include studies if they (1) the setting was using any sedative for endoscopy for an procedural sedation (2) the study compared dexmedetomidine with other sedative for sedative therapy and (3) the outcomes included satisfaction score and adverse events.
* Exclusion criteria We excluded studies if they (1) the number of sedative was different in two arms (2) did not report the specific results comparing dexmedetomidine with other sedatives.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two reviewers independently extract data, including outcomes of interests, demographics of the enrolled patients' population, inclusion and exclusion criteria for each study, the comparative drug used, the number of patients in each group, sedation target and posology.
Sampling Method: Non-Probability Sample
Enrollment: 6963 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects who experience desaturation | From first infusion of the sedative agent until awakening approximately up to 2 hours after the procedure.
  SaO2 < 94% for more than 10 seconds, RR<8, apneic episodes, face mask

SECONDARY OUTCOMES:
Number of subjects who experience Hypotension | From first infusion of the sedative agent until awakening approximately up to 2 hours after the procedure
  BP<90/50, decrease>20% or 10mmHg, MAP<60mmHg or MAP decrease>20%
Number of subjects who experience Bradycardia | From first infusion of the sedative agent until awakening approximately up to 2 hours after the procedure
  A heart rate of <50 beats per min, decrease > 15%

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0801043&StudyName=Sedation+Of+Adult+Patients+Undergoing+Gastrointestinal+Endoscopy%3A+A+Network+Meta-analysis